CLINICAL TRIAL: NCT05568680
Title: A Phase 1 Study of SynKIR-110, Autologous T Cells Transduced With Mesothelin KIR-CAR, in Subjects With Mesothelin-Expressing Advanced Ovarian Cancer, Cholangiocarcinoma, or Mesothelioma
Brief Title: SynKIR-110 for Mesothelin Expressing Ovarian Cancer, Cholangiocarcinoma or Mesothelioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Verismo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-101
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Cholangiocarcinoma Recurrent; Mesothelioma, Malignant
MeSH Terms: conditions — Ovarian Neoplasms; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SynKIR-110 (Experimental): Single dose gravity drip IV administration
  Interventions: Biological: SynKIR-110, Autologous T cells Transduced with Mesothelin KIR-CAR

INTERVENTIONS:
Biological: SynKIR-110, Autologous T cells Transduced with Mesothelin KIR-CAR — Autologous T cells Transduced with Mesothelin KIR-CAR

SUMMARY:
This first-in-human (FIH) trial is designed to assess the safety, feasibility, and potential activity of a single intravenous (IV) dose of SynKIR-110 administered to subjects with mesothelin-expressing advanced ovarian cancer, mesothelioma, and cholangiocarcinoma.

DETAILED DESCRIPTION:
This is a Phase 1, FIH, multicenter, open-label, dose-escalation pilot study of a single IV gravity drip infusion of SynKIR-110 in subjects with advanced, mesothelin-expressing tumors (ovarian cancer, primary peritoneal cancer, fallopian tube cancer, cholangiocarcinoma, or mesothelioma). Up to 42 subjects will be assessed to determine the safety and feasibility of treatment with SynKIR-110. Informed consent will be obtained from subjects prior to participation in this study.

The study includes an enrollment screening period (which includes pre-leukapheresis safety/eligibility and leukapheresis visits), treatment period (administration of non-myeloablative lymphodepleting chemotherapy followed by a single infusion of investigational product), and a 12-month follow-up period or until disease progression. Subjects will be followed for 12 months or until confirmed disease progression, whichever occurs first, at which point they will be invited to participate in a long-term safety follow-up study.

Up to 6 cohorts of 3 to 6 subjects per cohort will be treated to determine the safety and feasibility of treatment with SynKIR-110. Doses will be escalated following a standard 3 + 3 design until either an MTD or MFD is reached. An additional 6 to 9 subjects will be treated at the MTD/MFD to further assess safety and potential activity of SynKIR-110.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent or relapsed advanced ovarian cancer, primary peritoneal cancer, fallopian tube cancer, cholangiocarcinoma, or epithelial mesothelioma (pleural or peritoneal) after at least 1 prior line of systemic therapy for advanced disease
* Adult 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has at least 1 measurable lesion by iRECIST for ovarian cancer or cholangiocarcinoma or lesions measurable for mRECIST for mesothelioma.
* Satisfactory Blood coagulation parameters
* Satisfactory organ and bone marrow function

Exclusion Criteria:

* Active invasive cancers other than mesothelioma, cholangiocarcinoma, and ovarian unless surgically and medically cured without evidence of recurrent disease for 5 years.
* History of T or B cell malignancies or previous gene-engineered T cell therapies.
* Sarcomatoid/biphasic mesothelioma.
* Pulmonary exclusions
* Have acquired hereditary, congenital immunodeficiency or have recognized immunodeficiency disease
* Active hepatitis B, active hepatitis C, or any HIV infection at the time of screening
* Active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of SynKIR-110 | Up to 12 months
  * The incidence, frequency, and severity of TEAEs, incidence of AEs related to native mesothelin-expressing tissues, Incidence of CRS and/or neurologic toxicity
  * Frequency of subjects who pass screening to enrollment but do not receive SynKIR-110

SECONDARY OUTCOMES:
Define the maximum tolerated dose (MTD)/maximum feasible dose (MFD) of SynKIR-110 and to identify a recommended Phase 2 dose | Up to 12 months
  Define the MTD or MFD of SynKIR-110

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnson, PhD, Study Director — Verismo Therapeutics
Locations (4):
- United States (4):
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No